CLINICAL TRIAL: NCT05385926
Title: A Phase II Study: Safety and Efficacy of Combining Radiation Therapy With Immunotherapy and Chemotherapy in de Novo Metastatic Nasopharyngeal Carcinoma
Brief Title: Combining RT With Immunotherapy and Chemotherapy in Metastatic Nasopharyngeal Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, JIN JING, Head of Radiation Oncology, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JS2022-35
Record Dates: First submitted 2022-05-14; First posted 2022-05-23 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Metastatic Nasopharyngeal Cancer
Keywords: Metastatic Nasopharyngeal Cancer; PD-1; Radiotherapy; Chemotherapy
MeSH Terms: conditions — Nasopharyngeal Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RT group (Experimental)
  Interventions: Radiation: Radiotherapy

INTERVENTIONS:
Radiation: Radiotherapy — Patients who had complete response or partial response after at least 3 cycles (no more than 6 cycles) of chemotherapy combined with immunotherapy receive local radiotherapy 21 days. For those non-CR oligo-metastatic disease or symptomatic lesion, SBRT or conventional RT delivered. Maintenance therapy of immunotherapy for 2 years.

SUMMARY:
Incidences of de novo metastatic nasopharyngeal carcinoma range from 6% to 8% at the time of presentation. For the initial diagnosis of metastatic NPC, PD-1 plus chemotherapy yields a satisfactory outcome with1year PFS of 40%. Previous study demonstrated the benefit of adding radiotherapy to chemotherapy in metastatic NPC, however there is no evidence whether radiotherapy can further improve PFS based on chemotherapy plus PD-1 . The purpose of this study is to evaluate the safety and effectiveness of first-line immunochemotherapy combined with radiotherapy for initial diagnosed metastatic NPC.

ELIGIBILITY:
Inclusion Criteria:

* Age:18-75 years, male or female.
* ECOG 0-2
* Histologically or cytologically confirmed de novo metastatic nasopharyngeal carcinoma.(stage IVb, AJCC 8th)
* Complete response or partial response after at least 3 cycles (no more than 6 cycles) of chemotherapy combined with immunotherapy
* Measurable disease based on Response Evaluation Criteria In Solid Tumors (RECIST) 1.1.
* Adequate organ function.
* Patient has given written informed consent.

Exclusion Criteria:

* Unwilling or unable to provide informed consent
* Intolerance to radiotherapy or immunotherapy
* Patients who have head and neck radiotherapy history.
* previous or recent another malignancy, except for nonmelanoma skin cancer or cervical cancer in situ
* women in pregnancy, lactation period, or no pregnancy test 14 days before the first dose
* in other clinical trials within 30 days
* Patients with autoimmune disorder, including but not limited to systemic lupus erythematosus or multiple sclerosis;
* History of primary immunodeficiency
* History of active tuberculosis, drug-induced interstitial lung disease, or ≥ Grade 2 pulmonitis;
* Patients with human immunodeficiency virus (HIV) positive;
* Comorbidities that cannot be controlled by concomitant treatment, including but not limited to: ongoing or active infection, unexplained fever > 38.5°C (subjects with neoplastic fever are judged by the investigator to be included), symptomatic congestive heart failure ≥ Grade 2 according to New York Heart Association (NYHA) functional classification, LVEF (left ventricular ejection fraction) < 50%, hypertension poorly controlled by drugs, unstable angina, arrhythmia, active peptic ulcer disease or gastritis;
* not suitable for this study judged by researchers

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2022-05-05 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | 1year

SECONDARY OUTCOMES:
Overall survival (OS) | 1year
Objective response rate (ORR) | 4-8 weeks
Local-regional free survival (LRFS) | 1 year
Distant metastasis free survival (DMFS) | 1 year
Treatment-emergent adverse events | 1 year
  Incidence of treatment-emergent adverse events would be assessed based on the common toxicity criteria for adverse events version 5.0 (CTCAE v5.0)

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Center/National Clinical Research Center for Cancer/Cancer Hospital & Shenzhen Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Shenzhen, China

IPD SHARING:
Plan to Share IPD: No